CLINICAL TRIAL: NCT02652364
Title: Strong Ion Gap as Prognostic Indicator for Adult Patients Admitted With Shock to the Intensive Care Units
Status: Completed | Type: Observational
Sponsor: Singapore General Hospital (Other)
Collaborators: Changi General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2015/2423
Record Dates: First submitted 2016-01-07; First posted 2016-01-11 (Estimated); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Shock
MeSH Terms: conditions — Shock

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study evaluates if strong ion gap on admission or 24 hours after admission to critical care unit can predict 28 day outcome in patients admitted with shock due to any cause

DETAILED DESCRIPTION:
Metabolic acidosis is frequently found in patients with shock. Traditional methods of evaluating acid-base status can underestimate and even miss complex acid-base disorders particularly in the setting of hypoalbuminemia, hypo/hypernatraemia and hypo/hyperchloraemia .An alternative approach to acid-base balance, based on chemical and physical principles, and was proposed by Peter Stewart more than 30 years ago. Later in 1992 Figge and Fencl modified the strong ion difference, which corresponds with the net charge balance of all strong ions present in a given solution (the ''Fencl-Stewart'' approach). The strong ion gap (SIG) which corresponds with the difference between the apparent strong ion difference and the effective strong ion difference was proposed by Kellum. Compared to the Fencl- Stewart approach SIG has more accuracy and bedside practicality.

As the SIG is calculated from all known charged components of blood, it is considered the gold standard for the quantification of unmeasured anions. In contrast, the traditional anion gap calculation only factors in sodium, potassium, chloride and bicarbonate. In healthy humans, the SIG equals zero. In critically ill patients, a high SIG, defined as >2mEq/L, indicates the accumulation of unmeasured anions in blood as a cause of acidosis. The unmeasured anions include lactate, ketoacids, uraemic acids and toxins like ethylene glycol and methanol. Studies found that a higher SIG on admission to intensive care unit is associated with poorer outcomes, and has a role in prediction of outcome in septic patients. However this finding is not consistent.

In addition it was found that there is a significant difference in the threshold for SIG value associated with higher mortality. The abnormal SIG value in American studies are described around 5 mEq/l . However studies from Europe and Australia reported higher values in the range of 8-13 mEq/l. It is speculated that this difference is due to exogenous sources of unmeasured ions from gelatin based intravenous fluids used for resuscitation. Interestingly studies using gelatine- based fluids also failed to show a correlation between SIG and mortality. SIG values have not been published in critically ill Asian adult patients admitted to the Intensive Care Units (ICU) as yet. We aim to find the SIG for these patients in the hope that it will be useful for predicting outcome. Our hypothesis is that SIG is an independent predictor of outcomes in adult patient with shock.

We propose to conduct this prospective observational study in the surgical and medical ICUs of 2 hospitals in Singapore. (Singapore General Hospital and Changi General Hospital) We aim to enrol 112 of you admitted to the ICU with shock of any etiology. Shock is defined as persistence of arterial hypotension despite adequate volume resuscitation. Hypotension is defined as systolic pressure <90mmHg, Mean arterial pressure (MAP)<70 mmHg or drop in SBP >40 mmHg from baseline. 30ml/kg of fluid is considered as the threshold for adequate volume resuscitation.

The methodology of this observational study was approved by Sing health Institutional review Board, Singapore. We will include you if you have persistent hypotension despite adequate fluid resuscitation as defined above or if you require vasopressors or inotropes to maintain MAP above 65mmHg on admission.

We will exclude the conditions with acid base disturbance which are not amenable to using standard supportive care such as pre-existing chronic kidney disease stage 3 and above ( defined as estimated GFR<60 ml/min/1.73m2 ) and chronic liver failure.

Blood samples will be taken from indwelling intra-arterial catheters on admission and 24 hours after admission. Blood samples will be analyzed in the respective hospital laboratory for Arterial Blood Gas(ABG) analysis, electrolytes albumin and lactate levels in order to calculate the SIG.

All of you included in the study will be managed by the same group of critical care physician in accordance with pre-existing protocols in both ICUs to ensure that there will not be any major discrepancies among patients in terms of organ support and therapy. Haemodynamic support will be applied to reverse the hypotension and to correct peripheral perfusion abnormalities after optimal resuscitation. IV noradrenaline is the vasopressor of first choice followed by vasopressin and adrenaline.

Data collection-

Fluid resuscitation before ICU admission, SOFA and APACHE II score 24 hours after the admission, requirement for vasopressors, mechanical ventilation renal replacement therapy(RRT) ,duration of ICU stay, number of ventilator days, duration of vasopressor support, number of vasopressors used and the duration of RRT, 28 day outcome will be collected.

Calculation of SIG-

SIG will be calculated according to the following formulae;

1. SIG= SIDapp - SIDeff

   (SIDapp -Strong ion difference apparent; SIDeff - Strong ion difference effective)
2. SIDapp = ( Na++K++Ca2++Mg2+) - (Cl-+Lactate-)

   ( all concentrations in mEq/l)
3. SIDeff = 2.46 x 10-8 x Pco2/ 10-pH + [albumin] x ( 0.123xpH - 0.631) +[PO43-] x (0.309xpH -0.469)

(PCO2 is measured in mm Hg, albumin in g/L, and phosphate in mmol/L)

ELIGIBILITY:
Inclusion Criteria:

* Patient with any form of shock on admission to ICU

Exclusion Criteria:

* CKD stage 3 and above (GFR> 60)
* Chronic liver failure( Child's B grade and above)
* Patients who were already recruited for this study
* Patients expected to die within next 48 hrs upon admission

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with any form of shock on admission to ICU defined by those who require vasopressors or inotropes to maintain MAP > 65mmHg on admission
Sampling Method: Non-Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2015-10; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
mortality | 28 days

SECONDARY OUTCOMES:
Duration of ICU stay | 28 days
  number of days patient spent in ICU

CONTACTS AND LOCATIONS:
Locations (1):
- Singapore General Hospital, Singapore, Singapore

REFERENCES:
- [Result] Mecher C, Rackow EC, Astiz ME, Weil MH. Unaccounted for anion in metabolic acidosis during severe sepsis in humans. Crit Care Med. 1991 May;19(5):705-11. doi: 10.1097/00003246-199105000-00018. PMID 2026034
- [Result] Figge J, Mydosh T, Fencl V. Serum proteins and acid-base equilibria: a follow-up. J Lab Clin Med. 1992 Nov;120(5):713-9. PMID 1431499
- [Result] Figge J, Jabor A, Kazda A, Fencl V. Anion gap and hypoalbuminemia. Crit Care Med. 1998 Nov;26(11):1807-10. doi: 10.1097/00003246-199811000-00019. PMID 9824071
- [Result] Stewart PA. Modern quantitative acid-base chemistry. Can J Physiol Pharmacol. 1983 Dec;61(12):1444-61. doi: 10.1139/y83-207. PMID 6423247
- [Result] Kellum JA, Kramer DJ, Pinsky MR. Strong ion gap: a methodology for exploring unexplained anions. J Crit Care. 1995 Jun;10(2):51-5. doi: 10.1016/0883-9441(95)90016-0. PMID 7647842
- [Result] Gunnerson KJ. Clinical review: the meaning of acid-base abnormalities in the intensive care unit part I - epidemiology. Crit Care. 2005 Oct 5;9(5):508-16. doi: 10.1186/cc3796. Epub 2005 Aug 10. PMID 16277740
- [Result] Kellum JA. Closing the gap on unmeasured anions. Crit Care. 2003 Jun;7(3):219-20. doi: 10.1186/cc2189. Epub 2003 May 8. PMID 12793870
- [Result] Rutherford EJ, Morris JA Jr, Reed GW, Hall KS. Base deficit stratifies mortality and determines therapy. J Trauma. 1992 Sep;33(3):417-23. doi: 10.1097/00005373-199209000-00014. PMID 1404512
- [Result] Smith I, Kumar P, Molloy S, Rhodes A, Newman PJ, Grounds RM, Bennett ED. Base excess and lactate as prognostic indicators for patients admitted to intensive care. Intensive Care Med. 2001 Jan;27(1):74-83. doi: 10.1007/s001340051352. PMID 11280677
- [Result] Balasubramanyan N, Havens PL, Hoffman GM. Unmeasured anions identified by the Fencl-Stewart method predict mortality better than base excess, anion gap, and lactate in patients in the pediatric intensive care unit. Crit Care Med. 1999 Aug;27(8):1577-81. doi: 10.1097/00003246-199908000-00030. PMID 10470767
- [Result] Kaplan LJ, Kellum JA. Initial pH, base deficit, lactate, anion gap, strong ion difference, and strong ion gap predict outcome from major vascular injury. Crit Care Med. 2004 May;32(5):1120-4. doi: 10.1097/01.ccm.0000125517.28517.74. PMID 15190960
- [Result] Funk GC, Doberer D, Sterz F, Richling N, Kneidinger N, Lindner G, Schneeweiss B, Eisenburger P. The strong ion gap and outcome after cardiac arrest in patients treated with therapeutic hypothermia: a retrospective study. Intensive Care Med. 2009 Feb;35(2):232-9. doi: 10.1007/s00134-008-1315-1. Epub 2008 Oct 14. PMID 18853143
- [Result] Noritomi DT, Soriano FG, Kellum JA, Cappi SB, Biselli PJ, Liborio AB, Park M. Metabolic acidosis in patients with severe sepsis and septic shock: a longitudinal quantitative study. Crit Care Med. 2009 Oct;37(10):2733-9. doi: 10.1097/ccm.0b013e3181a59165. PMID 19885998
- [Result] Cusack RJ, Rhodes A, Lochhead P, Jordan B, Perry S, Ball JA, Grounds RM, Bennett ED. The strong ion gap does not have prognostic value in critically ill patients in a mixed medical/surgical adult ICU. Intensive Care Med. 2002 Jul;28(7):864-9. doi: 10.1007/s00134-002-1318-2. Epub 2002 Jun 14. PMID 12122523
- [Result] Rocktaeschel J, Morimatsu H, Uchino S, Bellomo R. Unmeasured anions in critically ill patients: can they predict mortality? Crit Care Med. 2003 Aug;31(8):2131-6. doi: 10.1097/01.CCM.0000079819.27515.8E. PMID 12973170
- [Result] Hayhoe M, Bellomo R, Liu G, McNicol L, Buxton B. The aetiology and pathogenesis of cardiopulmonary bypass-associated metabolic acidosis using polygeline pump prime. Intensive Care Med. 1999 Jul;25(7):680-5. doi: 10.1007/s001340050930. PMID 10470571
- [Result] Gunnerson KJ, Srisawat N, Kellum JA. Is there a difference between strong ion gap in healthy volunteers and intensive care unit patients? J Crit Care. 2010 Sep;25(3):520-4. doi: 10.1016/j.jcrc.2009.11.001. Epub 2009 Nov 25. PMID 19942401